CLINICAL TRIAL: NCT02357342
Title: Sirolimus Versus AntiVEGF for Wet AMD
Brief Title: Sirolimus Versus Anti-Vascular Endothelial Growth Factor (antiVEGF) for Wet AMD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RKM008
Record Dates: First submitted 2015-02-02; First posted 2015-02-06 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Sirolimus; Bevacizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus (Experimental): Intravitreal Sirolimus
  Interventions: Drug: Sirolimus
- Standard of Care intravitreal anti-VEGF (Active Comparator): anti-VEGF intravitreal injections
  Interventions: Drug: Standard of Care intravitreal injections of anti-VEGF

INTERVENTIONS:
Drug: Sirolimus — intravitreal injection
  Other Names: DE-109
  Arms: Sirolimus
Drug: Standard of Care intravitreal injections of anti-VEGF — intravitreal injections of anti-VEGF
  Other Names: avastin,bevacizumab, eylea, aflibercept,
  Arms: Standard of Care intravitreal anti-VEGF

SUMMARY:
Phase 2 clinical trial, single site, randomized, subject-masked study to determine safety and efficacy of intravitreal injections of Sirolimus in subjects with wet Age-Related Macular Degeneration (wet AMD) with persistent intraretinal or subretinal edema due to neovascular AMD despite previous AntiVEGF treatment.

DETAILED DESCRIPTION:
Forty subjects will be randomized to receive intravitreal Sirolimus or standard of care treatment in a 1:1 ratio. Over the course of the six month trial plus a 6 month optional extension, subjects will be evaluated monthly. Treatment with Sirolimus will be given at baseline, month 2 and month 4 with sham injections given at months 1, 3 and 5. For subjects in the extension Sirolimus will also be given at months 6, 8 and 10 with sham at month 7, 9, and 11. Subjects in the standard of care group will receive anti-VEGF injections or sham monthly. Retreatment criteria will be based upon continued subretinal edema, intraretinal edema or active chorioretinal neovascularization (CNV)

ELIGIBILITY:
Inclusion Criteria:

* best corrected visual acuity of 5-65, inclusive, in study eye
* presence of choroid neovascularization secondary to AMD
* persistent edema despite at least 3 previous intravitreal anti-VEGF injections in the past 5 months

Exclusion Criteria:

* greater than 100 micron decrease in central subfield thickness on Optical Coherence Topography (OCT) since last standard of care visit
* history of major ophthalmic surgery in the study eye in the past 3 months
* history of significant ocular disease or condition other than exudative AMD that may confound results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Raj K. Maturi, MD, PC
Locations (1):
- Raj K Maturi MD PC, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minturn RJ, Bracha P, Klein MJ, Chhablani J, Harless AM, Maturi RK. Intravitreal sirolimus for persistent, exudative age-related macular degeneration: a Pilot Study. Int J Retina Vitreous. 2021 Feb 16;7(1):11. doi: 10.1186/s40942-021-00281-0. PMID 33593448

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus: Intravitreal Sirolimus
  Sirolimus: intravitreal injection at baseline, month 2 and month 4. Sham injections at months 1, 3 and 5
- Standard of Care Intravitreal Anti-VEGF: Standard of Care intravitreal injections of either bevacizumab (1.25mg/0.05ml) or aflibercept (2mg/0.05ml). Bevacizumab injections were repeated at monthly intervals and aflibercept was given at baseline, month 2 and 4 and sham injections at months 1, 3 and 5. Subjects in this group continued the same drug they were on prior to joining the study.
Period: First 6 Months
Arm/Group | Sirolimus | Standard of Care Intravitreal Anti-VEGF
Started (15 subjects were still in study when it was extended; 13 subjects qualified for extension.) | 20 | 20
Completed | 18 (2 patients died. Neither deaths were study drug related.) | 20
Not Completed | 2 | 0
Not completed — Death | 2 | 0
Period: Extension Study
Arm/Group | Sirolimus | Standard of Care Intravitreal Anti-VEGF
Started | 4 | 9
Completed | 4 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Intravitreal antiVEGF: antiVEGF intravitreal injections
  Standard of Care intravitreal injections of antiVEGF: intravitreal injections of antiVEGF
- Total: Total of all reporting groups
Arm/Group | Sirolimus | Standard of Care Intravitreal antiVEGF | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 20 | 18 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 8 | 4 | 12
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Edema From Baseline to Month 6 Central Subfield Thickness ) on Heidelberg Optical Coherence Topography
Description: Change in edema from baseline to month 6 as measured by mean difference in microns of central subfield thickness on Heidelberg optical coherence topography in each treatment group
Time Frame: Baseline to 6 months
Measure: Mean (Full Range); unit: microns
Arm/Group | Sirolimus | Standard of Care Intravitreal Anti-VEGF
Number analyzed (Participants) | 18 | 20
microns | -30.0 [-136 to 76] | 7.5 [-113 to 128]

2. Primary Outcome: Visual Acuity
Description: number of subjects with gain of 0-4 letters of visual acuity
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus | Standard of Care Intravitreal Anti-VEGF
Number analyzed (Participants) | 18 | 20
Participants | 7 | 11

3. Secondary Outcome: Visual Acuity (Best Corrected Visual Acuity)
Description: number of subjects with gain of 5 or more letters of visual acuity
Time Frame: baseline to 6 months
Measure: Number (100% Confidence Interval); unit: participants
Arm/Group | Sirolimus | Standard of Care Intravitreal Anti-VEGF
Number analyzed (Participants) | 18 | 20
participants | 9 [0 to 10] | 9 [0 to 10]

ADVERSE EVENTS:
Time Frame: On or after baseline visit (Day 0) to on or before month 12 visit.
Arm/Group | Sirolimus | Standard of Care Intravitreal Anti-VEGF
All-Cause Mortality (participants affected / at risk) | 2/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 14/20 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus (N=20) | Standard of Care Intravitreal Anti-VEGF (N=20)
pulmonary embolism (Vascular disorders) | 1 (1) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
subretinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
central retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
anterior chamber inflammation (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sirolimus (N=20) | Standard of Care Intravitreal Anti-VEGF (N=20)
photopsia (Eye disorders) | 0 (0) | 1 (1)
underactive thyroid (Endocrine disorders) | 0 (0) | 1 (1)
unexplained vision Loss (Eye disorders) | 1 (1) | 0 (0)
intraretinal hemorrhage (Eye disorders) | 1 (1) | 1 (1)
hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
decreased visual acuity (Eye disorders) | 5 (5) | 1 (1)
angular blepharitis (Eye disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pre-cancerous lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
basal cell carcinoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dot hemorrhage (Eye disorders) | 1 (1) | 0 (0)
corneal irritation (Eye disorders) | 2 (2) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1/2 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Right radial artery hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Hypotic Respiratory failure (Reproductive system and breast disorders) | 1 (1) | 0 (0)
shingles (Nervous system disorders) | 0 (0) | 1 (1)
increased intraocular pressure (Eye disorders) | 2 (3) | 1 (1)
progressed posterior subcapsular cataract (Eye disorders) | 1 (2) | 0 (0)
progressed nuclear sclerotic cataract (Eye disorders) | 1 (1) | 0 (0)
Serous Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Subretinal Hemorrhage (Eye disorders) | 1 (1) | 1 (1)
choroidal neovascular membrane (Eye disorders) | 0 (0) | 1 (1)
intraretinal and subretinal fluid (Eye disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Worsening hypertension (Vascular disorders) | 0 (0) | 1 (1)
PRES syndrome (Nervous system disorders) | 0 (0) | 1 (1)
arthritis, left sholder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
Acute Chronic Hypoxic Respitory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diastolic Dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Acute Kidney Inury (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
uveitis (Eye disorders) | 1 (1) | 0 (0)
Posterior Synechiae (Eye disorders) | 1 (1) | 0 (0)
Endothelial Pigment (Eye disorders) | 1 (1) | 0 (0)
corneal edema (Eye disorders) | 1 (1) | 0 (0)
worsening anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
floaters (Eye disorders) | 0 (0) | 1 (1)
subconjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
recurrent subretinal hemorrhage (Eye disorders) | 1 (1) | 0 (0)
headache (right side of head) (General disorders) | 1 (2) | 0 (0)
eye pain following injection (Eye disorders) | 1 (2) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
parkinsons disease (Nervous system disorders) | 1 (1) | 0 (0)
pigment on lens surface (Eye disorders) | 1 (1) | 0 (0)
hemorrhage on optic nerve (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes